CLINICAL TRIAL: NCT00277173
Title: Improving Geriatric Drug Safety in Underserved Practices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: R21HS014867 (AHRQ)
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2006-01-16 (Estimated); Status verified 2006-01

CONDITIONS: Cardiovascular Diseases
Keywords: Medication Safety; Adverse Drug Events; Preventable Adverse Drug Events; Culture of Safety; Failure Modes and Effects Analysis; Teambuilding
MeSH Terms: conditions — Cardiovascular Diseases; Drug-Related Side Effects and Adverse Reactions

INTERVENTIONS:
Behavioral: Adoption of Crew Resource Management approach

SUMMARY:
The purpose of this study is to determine whether a CRM (adapted Crew Resource Management approach proven successful in aviation as well as some inpatient medical settings) intervention is effective for reducing medication errors among older adults in primary care settings.

DETAILED DESCRIPTION:
Adverse drug events (ADEs) are among the most common and serious medication use concerns among older patients in primary care practices, yet they are often preventable. This translational research into practice (TRIP) pilot study uses a randomized trial to evaluate the effect of a site-level intervention in a sample of practices in medically underserved communities within the Upstate New York Practice Based Research Network (UNYNET). These sites are located in rural and urban areas and include an over-sample of minority patients. The specific aims of this study are to:

1. Examine the feasibility of objectively assessing the impact of a CRM (adapted Crew Resource Management approach proven successful in aviation as well as some inpatient medical settings) intervention on reducing medication errors among geriatric patients in primary care settings; and
2. Assess office staff internalization and application of CRM principles for reducing geriatric medication errors in primary care settings by examining changes in safety attitude constructs achieved

   1. with a practice enhancement assistant (PEA) and
   2. without a PEA.

Outcomes measured for Aim #1 will be change in number, severity, consequence, and stage of process of preventable ADEs. Outcomes for Aim # 2 will be change in safety climate, teamwork climate, stress recognition, and working conditions.

Fifteen sites will be randomized into one of three intervention arms: usual care, CRM only, or CRM plus a PEA. A random sample of charts of older adults (aged >64) with cardiovascular disease will be reviewed for adverse drug events over prior-year periods at baseline and post-intervention endpoints. Participatory research methods will be used to assess provider- and staff-identified barriers to implementation. This study will test the feasibility of incorporating PEA's into the practice setting to improve geriatric medication safety. The information gathered will serve as a basis for an ongoing translational research program that will lead to an RO1 application.

ELIGIBILITY:
Practice Inclusion Criteria:

* Practice must located in Health Professional Shortage Area or Physician Scarcity Area.
* Practice must be a member of the Western New York Practice-Based Research Network

Practice Exclusion Criteria:

* None

Patient Inclusion Criteria (for chart review):

* Aged >64
* Cardiovascular disease
* Seen at the practice within the past year

Patient Exclusion Criteria (for chart review):

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4800
Dates: Start 2006-01

PRIMARY OUTCOMES:
Change in number of total and preventable ADEs.
Change in culture of safety

CONTACTS AND LOCATIONS:
Overall Officials: Gurdev Singh, MScEng. PhD., Principal Investigator — State University of New York at Buffalo
Locations (1):
- Family Medicine Research Institute, Buffalo, New York, United States